CLINICAL TRIAL: NCT02627846
Title: A Randomised Clinical Trial Comparing Endovenous Laser Ablation and Mechanochemical Ablation (ClariVein®) in the Management of Superficial Venous Insufficiency
Brief Title: Laser Ablation Versus Mechanochemical Ablation Trial
Acronym: LAMA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hull University Teaching Hospitals NHS Trust (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R1788
Record Dates: First submitted 2015-12-01; First posted 2015-12-11 (Estimated); Last update posted 2023-09-21 (Actual); Status verified 2023-08

CONDITIONS: Varicose Veins
MeSH Terms: conditions — Varicose Veins | interventions — Lidocaine; Sodium Bicarbonate; Sodium Tetradecyl Sulfate; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EndoVenous Laser Ablation (Active Comparator): EndoVenous Laser Ablation (EVLA) involves the delivery of laser light through a glass fibre placed into the lumen of a refluxing vein. This energy is converted into heat inducing a permanent, non-thrombotic occlusion.
  Interventions: Device: EVLA; Drug: Lidocaine with 1:200,000 epinephrine solution; Drug: Sodium Bicarbonate
- MechanoChemical Ablation (ClariVein®) (Active Comparator): Mechanochemical ablation (MOCA) is performed by a device called ClariVein® which is a long thin catheter that is passed up inside the vein, with a rotating wire that protrudes at an angle from the end when deployed. This is motorised via an electric motor in the handle and rotates at approximately 3500 revolutions per minute. In addition, liquid sclerotherapy is injected at the handle end by a syringe. This sclerotherapy liquid emerges from the end of the catheter and is present in the area of the rotating tip.
  Interventions: Device: ClariVein®; Drug: Lidocaine with 1:200,000 epinephrine solution; Drug: Sodium Tetradecyl Sulphate

INTERVENTIONS:
Device: EVLA — 1% Lidocaine with 1:200,000 epinephrine will be used for skin infiltration. The EVLA fibre is introduced into the vein using the Seldinger technique and its tip will be positioned under duplex ultrasound (DUS). Then tumescent anaesthetic, made of a solution of 100ml of 1% Lidocaine with 1:200,000 epinephrine in 900ml of 0.9% Sodium Chloride and buffered to pH 7.4 with 10ml of 8.4% Sodium Bicarbonate, will be infiltrated around the target axial vein under DUS using a spinal needle and a peristaltic pump. Following deployment of appropriate laser safety precautions, the laser energy will be delivered via the fibre. The wavelength used is 1470nm, with NeverTouch Gold-Tip fibre, at 10W power. This laser light energy is converted into heat inducing a permanent, non-thrombotic occlusion.
  Other Names: Endovenous Laser Ablation
  Arms: EndoVenous Laser Ablation
Device: ClariVein® — 1% Lidocaine with 1:200,000 epinephrine will be used for skin infiltration. MOCA is performed by a device called ClariVein® (Vascular Insights, UK) which is a long thin catheter that is passed up inside the vein, with a rotating wire that protrudes at an angle from the end when deployed. This is motorised via an electric motor in the handle and rotates at approximately 3500 revolutions per minute. In addition, liquid sclerotherapy is injected at the handle end by a syringe. This sclerotherapy liquid emerges from the end of the catheter and is present in the area of the rotating tip. The sclerosant will be Sodium Tetradecyl Sulphate (STS), marketed as Fibrovein. Concentration of 1.5% Fibrovein will be used, and maximum of 12ml.
  Other Names: Mechanochemical Ablation
  Arms: MechanoChemical Ablation (ClariVein®)
Drug: Lidocaine with 1:200,000 epinephrine solution — It is used as local anaesthetic given via subcutaneous injection, so that the skin is numb prior to the introduction of either endovenous laser ablation or mechenochemical ablation catheter. Typically 1-2ml is required.
  Other Names: Lignocaine with 1:200,000 adrenaline solution
Drug: Lidocaine with 1:200,000 epinephrine solution — 100ml of 1% lidocaine with 1:200,000 epinephrine is diluted into 900ml of 0.9% Sodium Chloride to make the tumescent anaesthetic solution, which is required when using endovenous laser ablation.
  Other Names: Lignocaine with 1:200,000 adrenaline solution
  Arms: EndoVenous Laser Ablation
Drug: Sodium Bicarbonate — 10ml of 8.4% Sodium Bicarbonate is added into the tumescent anaesthetic solution, to buffer the pH to 7.4. Tumescent anaesthetic solution is required when using endovenous laser ablation.
  Arms: EndoVenous Laser Ablation
Drug: Sodium Tetradecyl Sulphate — 1.5% of Sodium Tetradecyl Sulphate, marketed as Fibrovein, will be used with the mechanochemical ablation device (ClariVein®). This is a sclerosing agent with Manufacturer Authorisation, and it will be used unmodified. Intravenous injection causes intima inflammation and thrombus formation. This usually occludes the injected vein.
  Other Names: Fibrovein Solution for Injection
  Arms: MechanoChemical Ablation (ClariVein®)

SUMMARY:
A randomised clinical trial comparing endovenous laser ablation and mechanochemical ablation (ClariVein®) in the management of superficial venous insufficiency.

DETAILED DESCRIPTION:
Varicose veins, a very common problem in UK, may cause symptoms including pain, heaviness and itching in the lower legs. Overtime, bleeding and damage to surround soft tissues may develop, leading to venous ulcer which can be very painful, debilitating, difficult to heal and very expensive to treat.

Newer minimally invasive techniques are preformed using local anaesthetic. The recovery has been shown to be more rapid, due to less pain and disability when compared to open surgery. These techniques use either heat or a chemical/medicine injected inside the varicose veins to close them permanently. In 2013 National Institute of Health and Care Excellence (NICE) recommended that methods using heat such as endovenous laser ablation (EVLA) should be first choice as the chemical methods have been shown to have a significantly lower treatment success rates in closing varicose veins permanently. Chemical methods however do have their advantages, as they require far fewer injections of local anaesthetic than the heat methods and these injections can be a source of significant discomfort.

Since NICE guidelines, a new treatment technique known as mechanochemical ablation (MOCA) using ClariVein® has been developed. This device injects a chemical into the vein through a rotating hollow wire, which causes the vein to narrow and damages the lining of the vein, making the chemical more effective. This new treatment technique aims to match the success rates of the heat method, but with less pain since it avoids most of the local anaesthetic injections. Both treatments are currently used in the UK, however there is insufficient evidence as to whether one is better, or the same.

This trial will randomly allocate volunteer patients to have their varicose veins treated with either EVLA or MOCA. The investigators will assess a range of outcomes including pain scores, success rates, complications, quality-of-life and costs to see which, if any, of these treatments offer better results. Long term follow-ups will occur at 5 and 10 years.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 or over
* Symptomatic SVI which will likely benefit from treatment in the opinion of an experienced specialist and the participant
* Clinical grades C2-C6 on the CEAP system
* Superficial axial incompetence with proposed treatment lengths of at least 10cm
* Treatment with either endovenous laser ablation or mechanochemical ablation is technically feasible in the view of an experienced endovenous specialist
* Patient is willing to participate (including acceptance of randomisation to either treatment) and give valid, informed consent in the English language

Exclusion Criteria:

* One of the treatments is thought to be preferable by either the patient or an experienced endovenous specialist
* Unwilling or inability to comply with the requirements for follow-up visits
* Known allergy to medications or dressings used in the treatment
* Known right to left circulatory shunt
* Evidence of acute deep venous thrombosis or complete ipsilateral occlusion
* Pelvic vein insufficiency
* Active or recent thrombophlebitis (within 6 weeks)
* Impalpable foot pulses with an Ankle-Brachial Pressure Index of less than 0.8
* Pregnancy or breast feeding
* Active malignancy
* Immobility
* Involvement in other CTIMP trials within the last 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2023-09-04 (Actual)

PRIMARY OUTCOMES:
Intra-procedural Pain | Up to end of intervention
  Patient is asked immediately after the procedure of their level of pain experienced during the intervention; measured on a standardised visual analogue scale (VAS).
Technical Efficacy assessed by successful procedure defined as complete occlusion of the target vein segment. | At 1 year

SECONDARY OUTCOMES:
Aberdeen Varicose Vein Questionnaire (AVVQ) | 1 week, 6 weeks, 6 months, 1 year
  Disease Specific quality of life
Chronic Venous disease quality of life Questionnaire (CIVIQ-20) | 1 week, 6 weeks, 6 months, 1 year
  Disease Specific quality of life
VEnous INsufficiency Epidemiological and Economic Study to evaluate Quality of Life and Symptoms (VEINES-QOL/Sym) | 1 week, 6 weeks, 6 months, 1 year
  Disease Specific quality of life
Short Form 36 | 1 week, 6 weeks, 6 months, 1 year
  Generic quality of life
EuroQol (EQ5D) | 1 week, 6 weeks, 6 months, 1 year
  Generic quality of life
Post-procedural Pain | Throughout the first week after the procedure
  One week pain diary
Analgesia Use | 1 week
  One week analgesia diary
Bruising visual analogue scale | 1 week, 6 weeks, 6 months, 1 year
  Appreciation of the severity of bruising
Satisfactory visual analogue scale | 1 week, 6 weeks, 6 months, 1 year
  Satisfaction with treatment
Cosmesis visual analogue scale | 1 week, 6 weeks, 6 months, 1 year
  Satisfaction with cosmetic result from treatment
Recovery time | 1 week, 6 weeks, 6 months, 1 year
  Time taken to return to work (if employed) and daily activity
Complications | 1 week, 6 weeks, 6 months, 1 year
  Any numbness, persistent bruising, tenderness, skin loss/ulceration, lumpiness, development of thread, skin staining, wound infection, deep vein thrombosis, pulmonary embolus, stroke, loss of vision, damage to major artery, vein or nerve.
Recurrence of Varicose Veins | 1 week, 6 weeks, 6 months, 1 year
  Combination of history taking, clinical examination and duplex ultrasound assessment.
Disease Progression | 1 week, 6 weeks, 6 months, 1 year
  Comparison of clinical and duplex ultrasound findings between follow-ups.
Need for Further Treatment | 1 week, 6 weeks, 6 months, 1 year
  Comparison of clinical and duplex ultrasound findings between follow-ups is made and should there be failure of intervention or recurrence of varicose veins, there would be consultation between surgeon and patient to decide whether further intervention is required.

CONTACTS AND LOCATIONS:
Overall Officials: Ian Chetter, MBChB,MD,FRCS, Principal Investigator — Hull University Teaching Hospitals NHS Trust; Abduraheem Mohamed, MBBS,BSc,MRCS, Principal Investigator — Hull University Teaching Hospitals NHS Trust; Daniel Carradice, MBBS,MRCS,DipHE, Principal Investigator — Hull University Teaching Hospitals NHS Trust
Locations (1):
- Hull and East Yorkshire Hospitals NHS Trust, Hull, United Kingdom

REFERENCES:
- [Derived] Mohamed AH, Leung C, Wallace T, Smith G, Carradice D, Chetter I. A Randomized Controlled Trial of Endovenous Laser Ablation Versus Mechanochemical Ablation With ClariVein in the Management of Superficial Venous Incompetence (LAMA Trial). Ann Surg. 2021 Jun 1;273(6):e188-e195. doi: 10.1097/SLA.0000000000003749. PMID 31977509
- [Derived] Leung CC, Carradice D, Wallace T, Chetter IC. Endovenous laser ablation versus mechanochemical ablation with ClariVein((R)) in the management of superficial venous insufficiency (LAMA trial): study protocol for a randomised controlled trial. Trials. 2016 Aug 24;17(1):421. doi: 10.1186/s13063-016-1548-1. PMID 27552990
- See also: Abstract Link — https://www.ncbi.nlm.nih.gov/pubmed/27552990?dopt=Abstract
- See also: Abstract Link — https://trialsjournal.biomedcentral.com/articles/10.1186/s13063-016-1548-1
- See also: Abstract Link — https://journals.lww.com/annalsofsurgery/Abstract/2021/06000/A_Randomized_Controlled_Trial_of_Endovenous_Laser.30.aspx